CLINICAL TRIAL: NCT02688725
Title: Post-Mastectomy Surveillance to Detect Locally Recurrent Breast Cancer
Brief Title: Post-Mastectomy Surveillance to Detect Recurrence in Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 5617S-14
Record Dates: First submitted 2015-12-29; First posted 2016-02-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ultrasound (Experimental): post mastectomy ultrasound
  Interventions: Device: post mastectomy ultrasound

INTERVENTIONS:
Device: post mastectomy ultrasound — post mastectomy ultrasound

SUMMARY:
Currently, there is no standard recommendation for using imaging studies to check patients for breast cancer recurrence who have been treated with mastectomy. The investigator proposes performing in-office ultrasound examinations of these patients to determine if this would be helpful in identifying an expected 5-7% of patients with breast cancer recurrences following mastectomy.

DETAILED DESCRIPTION:
The investigator hypothesizes that surgeon-directed ultrasound is a feasible, accurate, and cost-effective strategy for local recurrence surveillance in breast cancer patients after mastectomy. Toward examining these hypotheses, the investigators propose the following Specific Aims:

Aim I: To determine the number of breast cancer recurrences following mastectomy detected by surgeon-performed ultrasound.

Aim II: To determine the sensitivity and specificity of surgeon-performed ultrasound for the detection of post-mastectomy breast cancer recurrence.

Aim III: To estimate the cost of performing surgeon-directed ultrasound for the detection of post-mastectomy breast cancer recurrence from the perspective of a third party payer relative to standard surveillance alone.

ELIGIBILITY:
Inclusion Criteria:

* must be ≥ 18 years of age.
* histologic diagnosis of invasive (ductal or lobular) or in situ (ductal) breast cancer (American Joint Committee on Cancer, 7th edition stage 0, I, II, III, or IV) -previously treated with mastectomy

Exclusion Criteria:

* pregnant or breast feeding.
* cannot tolerate lying supine for breast ultrasound examination.
* mastectomy for lobular carcinoma in situ, atypical ductal hyperplasia, or extensive microcalcifications in the absence of concurrent DCIS or invasive breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
To determine the number of breast cancer recurrences following mastectomy detected by surgeon-performed ultrasound. | 3 years
  To determine the number of breast cancer recurrences following mastectomy detected by surgeon-performed ultrasound during a three year trial period.

SECONDARY OUTCOMES:
The sensitivity of surgeon performed breast ultrasound to detect breast cancer recurrence after mastectomy will be measured. | 3 years
  Sensitivity measures the proportion of patients that have pathologically confirmed breast cancer recurrences that were correctly identified as such by surgeon performed ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Martinez, MD, MAS,FACS, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Regional Cancer Partnership, Everett, Washington, United States

IPD SHARING:
Plan to Share IPD: No